CLINICAL TRIAL: NCT03290118
Title: The Efficacy of Front-of-package Labelling Schemes: an Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Mary L'Abbe, Chair of the Department of Nutritional Sciences, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34393
Record Dates: First submitted 2017-09-08; First posted 2017-09-21 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Diet Modification; Cardiovascular Diseases; Nutrition
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traffic Light (Experimental): Participants in this group will be provided with a survey that shows the food and beverage packages with traffic light front of pack labels only.
  Intervention is the Nutrition Rating System - Traffic Light
  Interventions: Other: Nutrition Rating System - Traffic Light; Device: Smartphone application FoodFlip Device®
- Star System (Experimental): Participants in this group will be provided with a survey that shows the food and beverage packages with health star rating front of pack labels only.
  Intervention is the Nutrition Rating System - Health Star Rating
  Interventions: Other: Nutrition Rating System - Health Star; Device: Smartphone application FoodFlip Device®
- Warning Label (Experimental): Participants in this group will be provided with a survey that shows the food and beverage packages with warning front of pack labels only.
  Intervention is the Nutrition Rating System - Warning Labels
  Interventions: Other: Nutrition Rating System - Warning Label; Device: Smartphone application FoodFlip Device®
- Control (No Intervention): Participants in this group will be provided with a survey that shows the food and beverage packages without any front of pack labels.

INTERVENTIONS:
Other: Nutrition Rating System - Traffic Light — Behavioural: Nutrition Rating Systems (shown on the online survey and the mobile app) provide consumers with an interpretation of the healthfulness of a food or beverage, by indicating the levels (low=green, moderate=amber, high=red) of sodium, saturated fat and sugar in a product based on modified Food Standards Australia New Zealand (FSANZ) criteria.
  Arms: Traffic Light
Other: Nutrition Rating System - Health Star — Behavioural: Nutrition Rating Systems (shown on the online survey and the mobile app) provide consumers with an interpretation of the healthfulness of a food or beverage product by indicating the number of stars awarded to a product, from 0.5 to 5 stars, based on modified Food Standards Australia New Zealand (FSANZ) nutrient profiling criteria.
  Arms: Star System
Other: Nutrition Rating System - Warning Label — Behavioural: Nutrition Rating Systems (shown on the online survey and the mobile app) provide consumers with an interpretation of the healthfulness of a food or beverage product by indicating with a warning label products that are "high" in sodium, saturated fat and sugar, based on a percent daily value (%DV) greater than 15% for individual products and 30% for combination dishes.
  Arms: Warning Label
Device: Smartphone application FoodFlip Device® — This is embedded within each condition to inform and educate consumers about the labelling condition/intervention to which they are randomized. All participants are assigned to an app task to view 20 products and see the 'rating' these products would get according to their condition.
  Arms: Star System; Traffic Light; Warning Label

SUMMARY:
This is an online study that aims to test the effectiveness of Interpretative Nutrition Rating Systems (INRS) such as the Health Star Rating System (HSR or Star System), traffic light system and warning labels (high sodium, saturated fat and sugar) proposed by Health Canada. The study will incorporate the use of a Smartphone application (app), FoodFlip®, to help educate consumers on each INRS prior to their exposure on food packages.

ELIGIBILITY:
Inclusion Criteria:

* speak English as a primary language
* reside in Canada excluding the Northern Territories
* are 18 years or over
* provide informed consent
* do at least some of the household grocery shopping
* own a smartphone (version iPhone 3 or later or Android)
* are able to complete the survey on a minimum screen size of 9.7 inches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Comprehension task - ability to identify healthy products (survey measure) | 1 day (assessed immediately after app task and while viewing products with labelling system applied
  The participant's ability to identify the most healthy product in a group of 5 products in a task rating 5 products with varying levels of 'healthiness' according to modified FSANZ criteria. Question wording: Please rank these products in terms of healthiness where 1 is the"most healthy" and 5 is the "least healthy" cereal
Comprehension task - ability to identify unhealthy products (survey measure) | 1 day (assessed immediately after app task and while viewing products with labelling system applied
  The participant's ability to identify the least healthy product in a group of products in a group of 5 products in a task rating 5 products with varying levels of 'healthiness' according to modified FSANZ criteria. Question wording: Please rank these products in terms of healthiness where 1 is the"most healthy" and 5 is the "least healthy" cereal

SECONDARY OUTCOMES:
Comprehension task - ability to identify the overall 'healthiness' of a product (survey measure - Likert scale) | 1 day (assessed immediately after app task and while viewing products with labelling system applied
  The participant's ability to accurately rate a product as more or less healthy according to the type and amount of nutritional information on the product, using a 7 point Likert scale. Question wording: How healthy is this (product) for you?
Hypothetical purchasing of products (survey measure - Likert scale) | 1 day (assessed immediately after app task and while viewing products with labelling system applied
  The participant's perceived likelihood of purchasing a product according to the type and amount of nutritional information on the product, using a 7 point Likert scale.
  Question wording: Assume this product has a cost similar to other (product category). If you were shopping for (product), how likely would you be to purchase this one?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Vanderlee L, Franco-Arellano B, Ahmed M, Oh A, Lou W, L'Abbe MR. The efficacy of 'high in' warning labels, health star and traffic light front-of-package labelling: an online randomised control trial. Public Health Nutr. 2021 Jan;24(1):62-74. doi: 10.1017/S1368980020003213. Epub 2020 Oct 6. PMID 33019950
- [Derived] Ahmed M, Oh A, Vanderlee L, Franco-Arellano B, Schermel A, Lou W, L'Abbe MR. A randomized controlled trial examining consumers' perceptions and opinions on using different versions of a FoodFlip(c) smartphone application for delivery of nutrition information. Int J Behav Nutr Phys Act. 2020 Feb 12;17(1):22. doi: 10.1186/s12966-020-0923-1. PMID 32050996